CLINICAL TRIAL: NCT04492046
Title: The Effect of Complex Decongestive Applications on Lower Extremity Limb Volume in Patients With Lipedema
Brief Title: Complex Decongestive Applications in Patients With Lipedema
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gokhan Yazici, Principal Investigator, Gazi University
Other Study IDs: Lipedema
Record Dates: First submitted 2020-07-24; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Lipedema
Keywords: Lipedema; Manual lymph drainage; Complex Decongestive Physiotherapy
MeSH Terms: conditions — Lipedema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complex Decongestive physiotherapy: All participants included in the study were included in a treatment protocol consisting of Complex Decongestive physiotherapy.
  Interventions: Other: Manual Lymph Drainage; Other: Bandaging

INTERVENTIONS:
Other: Manual Lymph Drainage — Manual lymph drainage is an effective therapeutic method used in the conservative treatment of lipedema. The application was performed on both lower extremities for 45 minutes.
Other: Bandaging — Multilayered compression bandaging techniques have an assisting role in the further reduction of the volume of the limb and enhance the continuous pump mechanism via the active involvement of muscle pumps. All patients received bandages following Manual lymph drainage application.

SUMMARY:
Lipedema is a rare condition which almost exclusively affects women. The disease is characterized with bilateral, symmetric abnormal accumulation of subcutaneous fat and is often mistaken for simple obesity. In most patients, the hips, buttocks, thighs, knees, and lower legs are affected. Upper extremity involvement has been reported to be present in 80% patients. The hands and feet are never affected. The accumulation of subcutaneous fat and edema results in tenderness, sensitivity to touch and pressure and also pain. Patients also tend to bruise easily even after a minimal trauma. It has been reported that the complaint of pain increases with aging.There is no known cure for lipedema. However, conservative treatment with physiotherapy, manual lymph drainage and compression, also known as complex decongestive physiotherapy is used worldwide as a standard treatment regimen . The aim of this study is to investigate the effect of complex decongestive applications on lower extremity limb circumference and volume in patients with lipedema.

DETAILED DESCRIPTION:
All participants included in the study were included in a treatment protocol consisting of complex decongestive physiotherapy Each patient received;

1. 45 minutes of manual lymph drainage on both lower extremities,
2. Moisturisation of the lower extremities,
3. Bandage application

Alongside this routine, the patients were advised to exercise (walk) regularly every day.

This treatment routine was continued until the patients were discharged from the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the study
* Being 18-65 years old
* Having a diagnosis of lower extremity lipedema

Exclusion Criteria:

- Having edematous disease in the lower extremity such as lymphedema or chronic venous insufficiency

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients included in this study consisted of those who had a diagnosis of lipedema in the lower extremities, between the ages of 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Limb Volume | Change from Baseline limb volume at 6 weeks
  In measurement of limb volume, the perometer was used. The device measures limb volume via infrared light and it has been reported to be a quick and reliable method. The device has a square frame which is used to surround the perimeter of the limb. The limb interrupts the emitted infrared beams that would normally be sensed by the light-sensing diodes in the two planes. Thus two perpendicular diameter measurements of the limb for the measured segment are provided. The device estimates the opposite two sides based on an elliptical cross-section.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yazici, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volkan-Yazici M, Yazici G, Esmer M. The Effects of Complex Decongestive Physiotherapy Applications on Lower Extremity Circumference and Volume in Patients with Lipedema. Lymphat Res Biol. 2021 Feb;19(1):111-114. doi: 10.1089/lrb.2020.0080. Epub 2020 Oct 30. PMID 33124947